CLINICAL TRIAL: NCT02043418
Title: Outcome at 5 Years of Early Treated HIV Infected Infants on Antiretroviral Multi-therapy in the PEDIACAM ANRS12140 Project in Cameroon
Brief Title: Outcome at 5 Years of Early Treated HIV Infected Infants in the PEDIACAM Project
Acronym: PEDIACAM
Status: Active, not recruiting | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Centre Pasteur du Cameroun (Other); Centre Mère et Enfant de la Fondation Chantal Biya (Other); Centre Hospitalier D'essos (Other); Hospital General De Douala (Other); Institut Pasteur (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: ANRS 12140 -12225
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: HIV
Keywords: HIV; ARV; Pediatric; Cameroon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — a biobank (plasma / serum stored at -80 ° C) will be established
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- children VIH+: children infected with HIV
- Chlidren VIH-: uninfected children born from HIV-positive or HIV-negative mothers

SUMMARY:
This study aims to assess the long-term outcomes of children infected with HIV, having participated in the ANRS 12140 PediacamI study, in terms of: clinical and immunovirological response to ARV therapy, long-term ARV tolerance, and the impact of family environment and lifestyle on adherence to ARV treatment.

DETAILED DESCRIPTION:
The follow-up of HIV infected children is an important part of their access to antiretroviral drugs. This therapeutic follow-up has an impact on infant morbidity and mortality and remains challenging due to its complexity (multi-drug therapy), the use of galenic forms that are not well adapted to children, the risks of toxicity and their prolonged administration, and the evolution of this syndrome in the patients' parents. Currently, while access to ARV is being ameliorated for children in Sub-Saharan Africa, little information is available on medium to long-term evolution of early treated HIV infected infants on ARV treatment. In Cameroon, the PEDIACAM ANRS 12140 study assessed for a period of 2 years, the impact and feasibility of early ARV treatment in HIV infected children and their humoral responses to EPI vaccines.

This first study (PEDIACAM ANRS 12140) began in November 2007 and consisted of two phases. During the first phase all children born from HIV+ mothers in the maternity wards of the participating hospitals were invited to participate. For every infant born from an HIV+ mother, an infant born from an HIV- mother was matched. A total of 2052 pairs of infants were recruited and they were all followed up to the age of 14 weeks. All infants born from seropositive mothers had a PCR HIV diagnostic test at the age of 6 weeks.

The second phase began after the age of 14 weeks. It consisted of four groups of infants: a group of HIV+ infants born from HIV+ mothers and followed from birth (n=69); a group of HIV- infants born from HIV+ mothers and followed from birth (n=205); a control group including a subset of the HIV- children born from HIV- mothers that had been followed since birth (n=196); and a final group that was added at this phase including HIV+ children that had not been followed up since birth but who had been diagnosed before the age of 7 months at any of the trial sites (n=141). During this phase, children were followed up to the age of 2 years. During these two years (phase I and phase II) the following criteria were evaluated: feasibility of early ARV treatment in infants, treatment tolerance, efficacy and adherence, clinical and immuno-virological prognosis of HIV infection in infants, rate of MTCT according to prevention strategies and humoral response to vaccines,.

The prolongation to 5 years of follow-up of the children participating in Phase II of the study constitutes the present study, ANRS 12225 PEDIACAM II. This follow up includes HIV non-infected children and is a unique opportunity to describe the medium to long-term clinical and immunovirological prognosis of the HIV infection in children and to further identify factors associated with treatment failure.

This second part of PEDIACAM, is a prospective longitudinal, observational, national multi-centered study including two groups of infants: one group of HIV infected infants treated early, and one group of HIV non-infected infants (born to either HIV infected or HIV non-infected mothers). Participation in the study will be proposed to all the infants included in phase II of PEDIACAM ANRS 12140, if possible before the age of 2 years. Only children whose parents or legal guardians consent to this continuation of the follow-up will be included. The children participating in the study will be seen for consultation every 6 months until the last child included reaches the age of 5 years. In the course of each visit, a clinical examination will be carried out as well as a complete laboratory examination. Antiretroviral treatment will be in line with the national recommendations and guidelines.

Four hundred sixty (460) children including 148 HIV-infected and 312 HIV-uninfected have been included in ANRS 12225 - Pediacam II study. We hypothesize for the next three years follow up period a low rate of missing HIV-infected children (death or loss to follow up) of about 5% and 20% for HIV-uninfected children. With such hypothesis, we will have at the end of the study, information of 140 HIV-infected and 250 HIV-uninfected children for our analysis

This cohort will enable us to answer the questions that arise regarding the long-term outcomes of HIV infected children in terms of clinical prognosis and immunology, and the impact of family environment and lifestyle on ARV treatment adherence. It will also aid in structuring the follow-up of children treated with ARVs in Cameroon. Furthermore, this study will continue to observe the response to vaccines. It will enable the identification of possible failures in the vaccination program and will enable us to propose, if necessary, an adjustment of the vaccine calendar.

ELIGIBILITY:
Inclusion Criteria:

* infants having participated in the ANRS 12140 PEDIACAM study
* HIV+ or HIV-
* signed consent
* born from HIV+ mothers having received perinatal ARV therapy or not
* or HIV- mothers

Exclusion Criteria:

* unsigned consent form

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2007-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of clinical/biological events related to HIV infection | 5 years

SECONDARY OUTCOMES:
Number clinical/biological events grade 3 or higher and their potential relationship to ARV therapy, HIV infection or vaccines | 5 years
Emergence of genotypic mutations of viral resistance to treatment in infants with virologic failure | 5 years
  Virologic failure is defined by a value of viral load > 400 copies / ml measured by RT-PCR after 6 months of treatment
Survival of infants | 5 years
Age at switch to second line of ARV treatment | 5 years
  The duration of therapy without changes in treatment will also be monitored.
Clinical and immunovirological response to treatment | 5 years
  Success is defined as viral load < 400 copies/ml and a rise in CD4 count of at least 20% at 6 months of treatment, and no recorded drops in CD4 counts of more than 25%
Regularity of consultations and relationship of the person bringing the child to consultation. | 5 years
Death of parent or sibling | 5 years
Changes in living situation. | 5 years
  Changes of address and living space, separation of parents, changes of members of the family living with the infant (siblings, cousins, uncles, grandparents), transfer of the infant to public institutions or adoption, will all be monitored in the scheduled visits throughout the 5 year follow-up.
Communication of child's HIV status to family and community | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mathurin Tejiokem, Dr, Principal Investigator — Centre Pasteur du Cameroun; Albert Faye, Pr, Principal Investigator — Hopital Universitaire Robert-Debre
Locations (3):
- Cameroon (3):
  - Hôpital Laquintinie, Douala
  - Centre Hospitalier d'Essos, Yaoundé
  - Centre Mère et Enfant de la Fondation Chantal Biya, Yaoundé

REFERENCES:
- [Background] Kfutwah AK, Tejiokem MC, Ateba FN, Ndongo JA, Penda IC, Ngoupo PA, Tchendjou P, Chewa G, Boisier P, Rouzioux C, Warszawski J, Faye A; ANRS 12140-Pediacam Study Group. Seronegativation in early treated HIV-infected infants: frequency and potential implications on care and follow-up in a resource-limited country. J Acquir Immune Defic Syndr. 2011 Oct 1;58(2):e43-6. doi: 10.1097/QAI.0b013e31822d49f0. No abstract available. PMID 21921727
- [Background] Tejiokem MC, Faye A, Penda IC, Guemkam G, Ateba Ndongo F, Chewa G, Rekacewicz C, Rousset D, Kfutwah A, Boisier P, Warszawski J; ARNS 12140-PEDIACAM study group. Feasibility of early infant diagnosis of HIV in resource-limited settings: the ANRS 12140-PEDIACAM study in Cameroon. PLoS One. 2011;6(7):e21840. doi: 10.1371/journal.pone.0021840. Epub 2011 Jul 19. PMID 21818273
- [Result] Sofeu CL, Warszawski J, Ateba Ndongo F, Penda IC, Tetang Ndiang S, Guemkam G, Makwet N, Owona F, Kfutwah A, Tchendjou P, Texier G, Tchuente M, Faye A, Tejiokem MC; ANRS-PEDIACAM Study Group. Low birth weight in perinatally HIV-exposed uninfected infants: observations in urban settings in Cameroon. PLoS One. 2014 Apr 3;9(4):e93554. doi: 10.1371/journal.pone.0093554. eCollection 2014. PMID 24705410
- See also: Site of sponsor — http://anrs.fr